CLINICAL TRIAL: NCT02206724
Title: PROSPECTIVE EVALUATION OF STEREOTACTIC BODY RADIOTHERAPY FOR METASTATIC PROSTATE CANCER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll patients
Sponsor: Sharp HealthCare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140794
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STEREOTACTIC BODY RADIOTHERAPY (Experimental): STEREOTACTIC BODY RADIOTHERAPY to the prostate gland
  Interventions: Radiation: STEREOTACTIC BODY RADIOTHERAPY to the prostate gland

INTERVENTIONS:
Radiation: STEREOTACTIC BODY RADIOTHERAPY to the prostate gland

SUMMARY:
The investigators aim to test the safety and feasibility of prostate gland stereotactic body radiotherapy (SBRT) plus best systemic therapy in newly diagnosed metastatic prostate cancer.

DETAILED DESCRIPTION:
The investigators and other investigators have previously documented the safety and efficacy of definitive intent stereotactic body radiotherapy (SBRT) in the treatment of localized prostate cancer.

In the metastatic setting for multiple malignancies, improved survival rates and disease outcomes have been shown with definitive treatment of the primary disease site. This concept of "cytoreductive" surgery or decreasing the primary tumor burden is now considered the standard of care for metastatic colon, ovarian, renal cell, and some breast carcinomas (plus post-surgery irradiation).

With new guidelines and declining rates of PSA screening, the incidence of newly diagnosed metastatic prostate cancer is expected to increase. A recent population-based study has concluded significant improvements in the definitive treatment of the local prostate cancer in the stage IV setting with either radical prostatectomy or conventional prostate radiation treatments/brachytherapy. To our knowledge, one prospective phase II trial is currently accruing patients to best systemic therapy or best systemic therapy (BST) plus definitive treatment with either radical prostatectomy or conventionally fractionated radiation therapy

The investigators hypothesize that the addition of primary disease SBRT to best systemic therapy for newly diagnosed metastatic prostate cancer would be associated with an acceptable safety profile, quality of life, disease progression, and overall survival. The addition of SBRT to best systemic therapy is also expected to be better-received for stage IV patients (with relatively limited prognosis), vs. fully fractionated radiation therapy, brachytherapy, or radical prostatectomy. The above endpoints would initially be tested in a prospective phase II multi-institutional trial and in comparison with historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, adenocarcinoma of the prostate
* Clinical Stage T1b - T4, NX-0-1, M1
* Any Gleason score
* PSA<1000
* ECOG Performance Status 0-2
* No prior prostate radiation or other definitive therapy

Exclusion Criteria:

* Prior prostatectomy or cryotherapy of the prostate
* Prior radiotherapy to the prostate or lower pelvis
* Implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion
* Chemotherapy for a malignancy in the last 5 years
* History of an invasive malignancy (other than this prostate cancer, or basal or squamous skin cancers) in the last 5 years

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Radiation related toxicity | 5 years
  Radiation related toxicity as per history and physical, and 1 or several of Patient questionnaires:
  SF-12 questionnaire AUA questionnaire EPIC-26 questionnaire SHIM questionnaire Utilization of Sexual Medications/Devices questionnaire

SECONDARY OUTCOMES:
Feasibility | 3-4 years
  Feasibility in terms of accrual and practical treatment delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Sharp Healthcare, San Diego, California, United States